CLINICAL TRIAL: NCT03743688
Title: Kinetics of the Immune Response to Inactivated Influenza Vaccine in Healthy Adults
Acronym: KIRV
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Human Vaccines Project (Other)
Responsible Party: Principal Investigator, Buddy Creech, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 181619
Record Dates: First submitted 2018-10-31; First posted 2018-11-16 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Influenza; Influenza, Human; Vaccine Reaction; Influenza A; Influenza Type B; Influenza A H1N1; Influenza A H3N2
Keywords: Influenza Vaccine; Influenza
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and peripheral blood mononuclear cells will be collected and stored according to protocol for a variety of immune interrogations.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Influenza Vaccine Recipients (ccIIV-4): All participants will receive one dose of FDA-approved inactivated influenza vaccine (Flucelvax Quadrivalent) via intramuscular injection (0.5 mL) as part of their standard of care.
  Interventions: Biological: Influenza Vaccine Recipients

INTERVENTIONS:
Biological: Influenza Vaccine Recipients — 0.5 mL intramuscular injection
  Other Names: Flucelvax (ccIIV4)

SUMMARY:
The purpose of this study is to evaluate the body's immune response at different time points to an FDA-approved seasonal influenza vaccine. By better understanding the way the immune system responds to the influenza vaccine, the investigators can design more effective vaccines against influenza.

DETAILED DESCRIPTION:
This is an observational study of seasonal, cell-cultured inactivated influenza vaccine (cc-IIV4) in healthy males and non-pregnant females aged 18 to 45 years old, inclusive. This clinical study is designed to comprehensively evaluate the characteristics and kinetics of the immune response to influenza vaccine.

By developing a comprehensive understanding of the mechanisms by which the immune system responds to influenza vaccine, including innate immune system responses, the effect of early influenza exposures, and (eventually) the effect of potent adjuvants, the investigators will be better equipped to design more highly effective vaccines to conquer seasonal influenza and prevent influenza pandemics.

Data from this pilot observational study will guide the design of global studies addressing age-specific responses, the impact of sex and geography, and the role of adjuvants on influenza immunity.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study procedures.
* Are able to understand and comply with planned study procedures and be available for all study visits.
* Are males or non-pregnant females, 18-45 years of age, inclusive.
* Are in overall good health. (As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses that could affect the assessment of the immunogenicity of influenza vaccine.)
* Women of childbearing potential (not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful metal coil placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.) must use an acceptable contraception method (includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill")) from 30 days before vaccination until 30 days after vaccination.
* Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to vaccination.

Exclusion Criteria:

* Have an acute illness (an acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol) as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to vaccination.
* Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation.
* Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to vaccination.
* Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
* Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
* Have known hypersensitivity or allergy to components of cell-cultured influenza vaccine.
* Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
* Have a history of Guillain-Barre Syndrome.
* Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to vaccination.
* Received a licensed live vaccine within 30 days prior to vaccination, or plan to receive a licensed live vaccine within 30 days before or after vaccination.
* Received or plan to receive a licensed, inactivated vaccine within 14 days before or after vaccination.
* Received the 2018-2019 inactivated seasonal influenza vaccine prior to the study.
* Received immunoglobulin or other blood products (with exception of Rho D Ig) within 90 days prior to vaccination.
* Received an experimental agent within 30 days prior to vaccination or expect to receive an experimental agent during the study.
* Are participating or plan to participate in another clinical study with an interventional agent that will be received during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ten (10) individuals 18-45 years of age, 5 males and 5 non-pregnant females, who are in good health by history and meet all eligibility criteria, will be enrolled at one site participating in this study. The target population will reflect the community at large at the participating site.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Seroconversion (Hemagglutination (HAI) Assay) | 28 days after vaccination
  Percentage of subjects achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40 or a pre- vaccination HAI titer ≥1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) 28 days after vaccination.
Seroconverstion (Microneutralization (MN) Assay) | 28 days after vaccination
  Percentage of subjects achieving seroconversion (defined as either a pre-vaccination MN titer <1:10 and a post-vaccination MN titer ≥1:40 or a pre-vaccination MN titer ≥1:10 and a minimum four-fold rise in post-vaccination MN titer) 28 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Buddy Creech, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan.